CLINICAL TRIAL: NCT00411801
Title: A Blinded Non-inferiority Study to Compare Uniplas With Cryosupernatant Plasma in Thrombotic Thrombocytopenic Purpura (TTP)
Brief Title: Safety and Efficacy Study to Compare Uniplas With Cryosupernatant Plasma in Thrombotic Thrombocytopenic Purpura (TTP)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNI-108
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Thrombotic Thrombocytopenic Purpura (TTP)
Keywords: bleeding disorder; universal plasma; plasma; plasma exchange
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic; Hemostatic Disorders | interventions — Solvents

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uniplas (Experimental): Participants will receive Uniplas intravenously in 4 cycles of 7 to 9 days each for 1 month. The first cycle will consist of 1.5 plasma volume exchanges (= 75 mL/kg) for 3 consecutive days, followed by a minimum of 4 and a maximum of 6 daily single volume plasma exchanges (= 50 mL/kg). Subsequent treatment will depend upon the response of the participant to the first cycle, as assessed by a blinded assessor.
  Interventions: Biological: Uniplas
- Cryosupernatant plasma (Active Comparator): Participants will receive cryosupernatant plasma intravenously in 4 cycles of 7 to 9 days each for 1 month. The first cycle will consist of 1.5 plasma volume exchanges (= 75 mL/kg) for 3 consecutive days, followed by a minimum of 4 and a maximum of 6 daily single volume plasma exchanges (= 50 mL/kg). Subsequent treatment will depend upon the response of the participant to the first cycle, as assessed by a blinded assessor.
  Interventions: Biological: Cryosupernatant plasma

INTERVENTIONS:
Biological: Uniplas — Uniplas will be provided frozen in sterile plastic bags.
  Other Names: Blood group independent, universally applicable, prion-depleted, solvent/detergent treated, human pooled plasma
  Arms: Uniplas
Biological: Cryosupernatant plasma — Cryosupernatant plasma will be provided frozen in sterile plastic bags.
  Arms: Cryosupernatant plasma

SUMMARY:
Prior to the use of plasma products, thrombotic thrombocytopenic purpura (TTP) was usually a fatal condition. During plasma exchange therapy, patients need transfusion plasma that is blood group specific. Transfusing a patient with an incorrect blood group may have fatal consequences. Uniplas is a universally applicable human plasma, which can be administered irrespective of the patient's blood group. This study will test the safety and efficacy of Uniplas in comparison to cryosupernatant plasma in treatment of patients with TTP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above.
* Definite diagnosis of acute thrombotic thrombocytopenic purpura (TTP).
* Thrombocytopenia.
* Diagnostic signs of microangiopathic hemolytic anemia.

Exclusion Criteria:

* Congenital thrombotic microangiopathies.
* Alternative secondary cause for microangiopathy.
* Co-morbid illness limiting life expectancy to less than 3 months independent of TTP.
* Patients known to be HIV positive.
* Patients known to have lupus.
* Refusal to accept blood products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in (log) platelet count 1 month after treatment initiation | Baseline to Month 1
  Log platelet count was reported in units, where 1 unit = 10^9/L platelets.

SECONDARY OUTCOMES:
Percentage of participants who died at 1 and 3 months after treatment initiation | Baseline to Month 3
Percentage of participants with a complete response (CR), a partial response (PR), a non-response (NR), or a transient response (TR) after the first treatment cycle and at 1 month | Baseline to Month 1
  A CR was defined as a platelet count > 150 x 10^9/L on 2 consecutive days, and a decrease of lactate dehydrogenase (LDH) to within 1.25 times the upper limit of the normal range, and a resolution of previous neurological symptoms, and no new neurological symptoms. A PR was defined as at least a 2-fold increase in platelet count from baseline which is > 50 x 10^9/L. A NR was defined as a < 2-fold increase in platelet count, or a platelet count < 50 x 10^9/L, or severe red blood cell (RBC) fragmentation, or the development of new neurological symptoms, or no improvement in neurological status as defined by the level of consciousness. A TR was defined as achievement of a complete or partial response which then deteriorated, defined by a 50% decrease in peak platelet count, or neurological deterioration, or a 100% increase in nadir LDH level, or severe RBC fragmentation.
Total volume of plasma exchange fluid administered during treatment cycles up to 1 month | Baseline to Month 1
Time to reach maximum platelet count | Baseline to the end of the study (up to 7 months)
  Platelet count was reported in units, where 1 unit = 10^9/L platelets.
Best clinical response (complete response [CR], partial response [PR], non-response [NR], transient response [TR]) during the study | Baseline to the end of the study (up to 7 months)
  The percentage of participants with a CR, PR, NR, or TR, as their best clinical response during the study, is reported. A CR was defined as a platelet count > 150 x 10^9/L on 2 consecutive days, and a decrease of lactate dehydrogenase (LDH) to within 1.25 times the upper limit of the normal range, and a resolution of previous neurological symptoms, and no new neurological symptoms. A PR was defined as at least a 2-fold increase in platelet count from baseline which is > 50 x 10^9/L. A NR was defined as a < 2-fold increase in platelet count, or a platelet count < 50 x 10^9/L, or severe red blood cell (RBC) fragmentation, or the development of new neurological symptoms, or no improvement in neurological status as defined by the level of consciousness. A TR was defined as achievement of a complete or partial response which then deteriorated, defined by a 50% decrease in peak platelet count, or neurological deterioration, or a 100% increase in nadir LDH level, or severe RBC fragmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Frenzel, M.D., Study Director — Octapharma
Locations (1):
- Contact Octapharma for Facility Details, Centreville, Virginia, United States